CLINICAL TRIAL: NCT06170853
Title: The Effect of Exercise with AR Glasses on Metabolic Parameters and Anthropometric Measurements in Obese Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Harun Özbey, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023/198
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Childhood Obesity
Keywords: Childhood Obesity; Adolescent; Metabolic Parameters; Augmented Reality Glasses; Anthropometric Values
MeSH Terms: conditions — Pediatric Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Augmented reality glasses group (Experimental): Three days a week (12 weeks in total), each session will be 60 minutes in total, and moderate exercise will be done with AR glasses.
  Interventions: Other: Exercise with augmented reality glasses
- Control group (No Intervention): No intervention/application will be made to the children who will be included in the control group.

INTERVENTIONS:
Other: Exercise with augmented reality glasses — Three days a week (12 weeks in total), each session will be 60 minutes in total, and moderate exercise will be done with AR glasses.
  Arms: Augmented reality glasses group

SUMMARY:
This study was planned as a randomized controlled experimental study to determine the effect of exercise with Augmented Reality Goggles (AR) on metabolic parameters and anthropometric measurement values in obese children aged 10-19 years. The study will be conducted with children diagnosed with obesity between the ages of 10-19 years who are followed up in the Pediatric Endocrinology Outpatient Clinic of Erciyes University Health Application and Research Center Fevzi Mercan-Mustafa Eraslan Children's Hospital. According to the sample calculation, a total of 20 obese children aged 10-19 years (AR exercise group=10 and control group=10) will be included in the sample of the study. The data of the study will be collected using the Descriptive Characteristics Form for Obese Children and Their Families, Serum and Urine Biochemistry Values Form, Anthropometric Measurement Values Form, Augmented Reality Goggles, Body Composition Analyzer, Caliper, Tape Measure and Digital Height and Weight Measurement Device. Ethics committee permission was obtained from "Erciyes University Clinical Research Ethics Committee" and institutional permission was obtained from ERU Health Practice and Research Center Mustafa Eraslan Fevzi Mercan Children's Hospital. Hypothesis tests, correlation and regression analyzes will be applied according to the suitability of the data for normal distribution. As a result of the study, it is expected that exercise application with AR glasses will improve metabolic parameters and anthropometric measurement values in obese children.

DETAILED DESCRIPTION:
Obesity, which is one of the major health problems in both developed and developing countries today, is a health problem that occurs with an increase in adipose tissue when energy intake is higher than energy consumption and can cause social, psychological and serious medical problems. If current trends continue, it is reported that 70 million children may be obese and overweight by 2025 and obesity will be a leading health problem. Childhood obesity increases in the first year of life, between 5-6 years of age and during puberty. 1/3 of obese children and 80% of obese adolescents remain obese when they reach adulthood. On the other hand, it is known that 30% of adult obesity cases date back to childhood. It has been reported that obesity affects 10.9-20.0% of all children and adolescents. In a study involving 5206 school-age children (mean age 8.6±1.2 years, 50.2% boys) from seven European countries (Turkey, Bulgaria, Romania, Lithuania, Germany, Italy and the Netherlands), it was reported that the prevalence of obesity in Turkish children was 7.7%, the second highest in Europe after Romania. Obesity in childhood has many medical adverse effects on children. Obesity may cause problems such as rapid growth, early menstruation, increase in blood lipids, increase in heart rate and heart rate volume, fatty liver, impaired sugar metabolism, hypertension, increase in white adipose tissue, increase in serum irisin, myonectin, triglyceride, total cholesterol and leptin levels and decrease in omentin-1 levels. In studies conducted in obese and healthy children, it was found that triglyceride, total cholesterol, irisin, low density lipoprotein (LDL-C) and leptin concentrations were higher in obese children compared to healthy children and omentin-1 levels were lower. Considering that childhood obesity continues into adulthood and brings many problems, the importance of combating obesity in this period is clearly seen. Reducing calorie intake, increasing exercise and providing psychosocial support are very important in the fight against obesity. While exercise constitutes a part of the standard treatment of obesity, it has been reported to be more effective than diet because it increases energy expenditure. In studies conducted in obese children, it was found that planned and long-term moderate exercise increased serum irisin, myonectin, omentin-1 and HDL concentrations and decreased serum leptin, triglyceride, total cholesterol and LDL concentrations. It has also been reported that exercise reduces metabolic and cardiovascular complications and improves body composition, cardiovascular health and mental health. Despite the numerous benefits of exercise, it has been reported that regular exercise habits are low in obese children. It has been reported that obese children cannot exercise regularly due to reasons such as low motivation, parents' inability to spare time to spend time with their children, children who are overwhelmed between courses/courses in the exam marathon with career anxiety, lack of emotional support and inability to give up existing habits. In this direction, exercise that requires continuity in the management of childhood obesity can be made dynamic for obese children by using different approaches. Therefore, it is thought that structured exercise with augmented reality glasses (AR) that can respond to the reactions of the obese child will be more dynamic, improve metabolic and anthropometric values and prevent macrovascular complications that may develop in obese children. This study was planned as a randomized controlled experimental study to determine the effect of exercise with AR glasses on metabolic parameters and anthropometric measurement values in obese children aged 10-19 years.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 10-19,
* Having been diagnosed with childhood obesity at least six months ago,
* Do not have any other chronic disease,
* No psychiatric diagnosis,
* No orthopedic problems,
* Able to read and write
* Can speak Turkish,
* No mental, physical or neurological disability,
* Residing in the province where the research will be conducted,
* Children and children with parental consent to participate in the study will be included in the study.

Exclusion Criteria:

-

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in serum leptin levels | Change in average serum leptin over 12-week sessions
  Serum leptin of children with type 1 diabetes before, during, after exercise and during the control session.
Change in serum irisin levels | Change in average serum irisin over 12-week sessions
  Serum irisin of children with type 1 diabetes before, during, after exercise and during the control session.
Change in body mass index | Change in average body mass index over 12-week sessions
  Average body mass index values of children with obesity before, during, after exercise and during the control session.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Bayat, PhD, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No